CLINICAL TRIAL: NCT01906905
Title: A Comparative Trial of TMS Approaches to Treating Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor Colleen Loo, Black Dog Institute, The Prince of Wales Hospital, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HC13053
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transcranial Magnetic Stimulation (Active Comparator): Active TMS (1)
  Interventions: Device: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation 2 (Active Comparator): Active TMS (2)
  Interventions: Device: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation 3 (Active Comparator): Active TMS (3)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
Trancranial Magnetic Stimulation (TMS) is a non-drug and non-invasive treatment for depression and has been investigated for the treatment of psychiatric illness for over 15 years. There is now established evidence indicating TMS is an effective treatment for depression. However, the effectiveness of TMS varies between people, thus requiring further research to investigate its optimal application. Investigators want to compare the effectiveness of different forms of TMS, given with differing stimulation settings to the right or left side of the brain that has been associated with depression. This could potentially help clinicians in the future to improve the prescription of TMS as a treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. DSM-IV diagnosis of current Major Depressive Episode.
3. MADRS score of 20 or more.
4. Able to give informed consent.

Exclusion Criteria:

1. DSM-IV psychotic disorder.
2. Drug or alcohol abuse or dependence (preceding 3 months).
3. Inadequate response to ECT (current episode of depression).
4. Rapid clinical response required, e.g. high suicide risk.
5. Significant neurological disorder, which may pose increased risks with TMS, e.g., epilepsy.
6. Metal in the cranium, skull defects, pacemaker, cochlear implant, medication pump or other electronic device.
7. Pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale(MADRS) | Participants will be assessed for changes for duration of trial, an expected average of 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MB.BS. (Hons), FRANZCP, MD., Principal Investigator — Black Dog Institute, University of New South Wales
Locations (1):
- Black Dog Institute, University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Loo CK, Mitchell PB. A review of the efficacy of transcranial magnetic stimulation (TMS) treatment for depression, and current and future strategies to optimize efficacy. J Affect Disord. 2005 Nov;88(3):255-67. doi: 10.1016/j.jad.2005.08.001. Epub 2005 Sep 2. PMID 16139895
- [Background] Andrews G, Henderson S, Hall W. Prevalence, comorbidity, disability and service utilisation. Overview of the Australian National Mental Health Survey. Br J Psychiatry. 2001 Feb;178:145-53. doi: 10.1192/bjp.178.2.145. PMID 11157427
- [Background] Dodick DW, Schembri CT, Helmuth M, Aurora SK. Transcranial magnetic stimulation for migraine: a safety review. Headache. 2010 Jul;50(7):1153-63. doi: 10.1111/j.1526-4610.2010.01697.x. Epub 2010 Jun 10. PMID 20553334
- [Background] Kupfer DJ, Frank E. The interaction of drug- and psychotherapy in the long-term treatment of depression. J Affect Disord. 2001 Jan;62(1-2):131-7. doi: 10.1016/s0165-0327(00)00357-8. PMID 11172880
- [Background] Sachdev PS, McBride R, Loo C, Mitchell PM, Malhi GS, Croker V. Effects of different frequencies of transcranial magnetic stimulation (TMS) on the forced swim test model of depression in rats. Biol Psychiatry. 2002 Mar 15;51(6):474-9. doi: 10.1016/s0006-3223(01)01298-7. PMID 11922882
- [Background] Slade T, Johnston A, Oakley Browne MA, Andrews G, Whiteford H. 2007 National Survey of Mental Health and Wellbeing: methods and key findings. Aust N Z J Psychiatry. 2009 Jul;43(7):594-605. doi: 10.1080/00048670902970882. PMID 19530016
- [Result] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Result] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Result] Nahas Z, Bohning DE, Molloy MA, Oustz JA, Risch SC, George MS. Safety and feasibility of repetitive transcranial magnetic stimulation in the treatment of anxious depression in pregnancy: a case report. J Clin Psychiatry. 1999 Jan;60(1):50-2. doi: 10.4088/jcp.v60n0111. PMID 10074879
- [Result] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Result] Padberg F, Zwanzger P, Keck ME, Kathmann N, Mikhaiel P, Ella R, Rupprecht P, Thoma H, Hampel H, Toschi N, Moller HJ. Repetitive transcranial magnetic stimulation (rTMS) in major depression: relation between efficacy and stimulation intensity. Neuropsychopharmacology. 2002 Oct;27(4):638-45. doi: 10.1016/S0893-133X(02)00338-X. PMID 12377400
- [Result] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Result] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Result] Slotema CW, Blom JD, Hoek HW, Sommer IE. Should we expand the toolbox of psychiatric treatment methods to include Repetitive Transcranial Magnetic Stimulation (rTMS)? A meta-analysis of the efficacy of rTMS in psychiatric disorders. J Clin Psychiatry. 2010 Jul;71(7):873-84. doi: 10.4088/JCP.08m04872gre. Epub 2010 Mar 9. PMID 20361902
- [Result] Speer AM, Benson BE, Kimbrell TK, Wassermann EM, Willis MW, Herscovitch P, Post RM. Opposite effects of high and low frequency rTMS on mood in depressed patients: relationship to baseline cerebral activity on PET. J Affect Disord. 2009 Jun;115(3):386-94. doi: 10.1016/j.jad.2008.10.006. Epub 2008 Nov 22. PMID 19027962
- [Result] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057